CLINICAL TRIAL: NCT02592681
Title: Comparison of the Prophylactic Effect Between Acupuncture and Acupressure on Menstrual Migraine
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Western University, Canada (Other)
Responsible Party: Principal Investigator, Alan Salmoni, Professor, Western University, Canada
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: WesternUCanada-acu
Record Dates: First submitted 2015-10-27; First posted 2015-10-30 (Estimated); Last update posted 2015-10-30 (Estimated); Status verified 2015-10

CONDITIONS: Menstrual Migraine
Keywords: menstrual migraine; acupuncture; acupressure
MeSH Terms: interventions — Acupressure

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- verum acupuncture (Experimental): Participants will receive real needle insertion. The needles will be left in the acupoint for 20 min, with a manual rotation at a ten-min interval. Primary acupoints used in the verum acupuncture group will be: LR3 (Taichong), LI4 (Hegu), SP6 (Sanyinjiao), GB20 (Fengchi). Extra acupoints will be selected based on TCM pattern are GB41 (Zulinqi), SP10 (Xuehai), KI3 (Taixi), or LR2 (Xingjian).
  Interventions: Procedure: verum acupuncture
- acupressure (Active Comparator): Acupressure will be applied on all the corresponding acupoints described in the acupuncture group. Duration of each session will be 15 min.
  Interventions: Procedure: acupressure
- control acupuncture (Sham Comparator): The number, duration, and frequency of the sessions will be the same as for the verum acupuncture group. The points chosen will be: LR7 (Xiguan), GB35 (Yangjiao), LI12 (Zhouliao), M-BW-1 (Dingchuan).
  Interventions: Procedure: control acupuncture

INTERVENTIONS:
Procedure: verum acupuncture — Participants will receive real needle insertion. Sterile needles will be used on all acupoints. The depth of insertion will vary from 15 mm to 20 mm depending on the exact locations. An initial manual stimulation will be given at insertion by rotation methods to produce a specific sensation described as "de-qi" in TCM. Then the needles will be left in the acupoint for 20 min, with a manual rotation at 4-8 Hz and an amplitude of approximately 0.5-2 rotations at a ten-min interval to maintain the sensation of "de-qi". Primary acupoints used in the verum acupuncture group will be: LR3 (Taichong), LI4 (Hegu), SP6 (Sanyinjiao), GB20 (Fengchi). Extra acupoints will be selected based on TCM pattern are GB41 (Zulinqi), SP10 (Xuehai), KI3 (Taixi), or LR2 (Xingjian).
  Arms: verum acupuncture
Procedure: acupressure — The acupoints and the number of the sessions will be exactly the same as for the verum acupuncture group. Acupressure will be applied on all the corresponding acupoints described in the acupuncture group. Finger pressure will be applied to each acupoint for eight seconds followed by two-seconds rest, repeated for 3 min. The strength of the pressure depends on individual participant's sensation of "de-qi". Duration of each session will be 15 min.
  Arms: acupressure
Procedure: control acupuncture — The number, duration, and frequency of the sessions will be the same as for the verum acupuncture group. Sterile needles will be used on acupoints that have no therapeutic effect on either menstruation or migraines, based on the acupuncture text books and acupuncture research literature. The points chosen will be: LR7 (Xiguan), GB35 (Yangjiao), LI12 (Zhouliao), M-BW-1 (Dingchuan). The depth of needle insertion will be as superficial as 3 mm, and without manual rotation, in order to minimize stimulation of the needle.
  Arms: control acupuncture

SUMMARY:
This study is designed to make comparisons between acupuncture and acupressure for preventing menstrual migraine (MM). Whether acupuncture is superior to acupressure is the most interesting point of this study. First of all, females will be screened for eligibility. Then, all participants who meet the inclusion criteria will be asked to keep a headache migraine diary for three months as baseline data. The diaries will then be collected before the first treatment. Then, all the participants will receive the corresponding interventions on the eighth, fifth and second days before the estimated first day of menstruation (determined individually from the diaries) in each month for three months (menstrual cycle), making a total of nine treatment sessions. After the whole treatments, there will be a three-month follow-up period. All the participants will be asked to complete the headache diaries every month from baseline to the end of the study. The diaries recording data from the fourth to the ninth month will then be collected at the end of the ninth month for the second time indicating the end of the study for the participants. In case of an acute migraine attack, participants will not be restricted from using "normal" medications.

DETAILED DESCRIPTION:
First of all, the females who are interested in this study will have an appointment with the researcher to decide their eligibility according to the inclusion and exclusion criteria. If eligible, participants will then sign a consent form.

Then, all participants who meet the inclusion criteria will be asked to keep a headache diary in which they will record the date of any migraine attacks, starting and ending time point of each migraine attack, drug usage (doses and type), average migraine pain on a 10-point VAS, and days of menstruation, during a three-month period (three menstrual cycles). The diaries will be collected by the researcher at the end of the third month and the traditional Chinese medicine (TCM) patterns of MM of the participants will be diagnosed then according to answering a few symptom related questions. In addition, times/dates for treatments will be scheduled.

Upon arrival at the exercise lab, Room 4115 inside Thames Hall in Western University on the first treatment day (the eighth day before the estimated first day of menstruation), participants will be asked to sit and relax for 1-2 min. Then they will be asked to lie down in a prone position receive corresponding interventions by the acupuncturist.

In the verum acupuncture group, participants will receive real needle insertion. Sterile needles (0.18 mm in diameter and 30 mm in length, DONGBANG Needle, Korea) will be used on all acupoints. The depth of insertion will vary from 15 mm to 20 mm depending on the exact locations. An initial manual stimulation will be given at insertion by rotation methods to produce a specific sensation described as "de-qi" in TCM (a sensation perceived by the acupuncture receivers as numbness, fullness, and sometimes soreness around the point. Then the needles will be left in the acupoint for 20 min, with a manual rotation at 4-8 Hz and an amplitude of approximately 0.5-2 rotations at a ten-min interval to maintain the sensation of "de-qi".

Primary acupoints used in the verum acupuncture group will be: LR3 (Taichong), LI4 (Hegu), SP6 (Sanyinjiao), GB20 (Fengchi). They are selected according to several previous relevant clinical studies. Extra acupoints will be selected based on TCM pattern. If it is due to qi stagnation, GB41 (Zulinqi) will be added. If it is due to blood stasis, SP10 (Xuehai) will be added. If it is due to Liver and Kidney yin deficiency, KI3 (Taixi) will be added. If it is due to Liver fire, LR2 (Xingjian) will be added. The exact localizations of these acupoints are described in a textbook. All these points will be applied bilaterally unless there are explicit reasons for not doing so being described in details.

In the acupressure group the acupoints and the number of the sessions will be exactly the same as for the verum acupuncture group. Acupressure will be applied on all the corresponding acupoints described in the acupuncture group. Finger pressure will be applied to each acupoint for eight seconds followed by two-seconds rest, repeated for 3 min. The strength of the pressure depends on individual participant's sensation of "de-qi". Duration of each session will be 15 min.

In the control acupuncture group, the number, duration, and frequency of the sessions will be the same as for the verum acupuncture group. Sterile needles (0.18 mm in diameter and 15 mm in length, DONGBANG Needle, Korea) will be used on acupoints that have no therapeutic effect on either menstruation or migraines, based on the acupuncture text books and acupuncture research literature. The points chosen will be: LR7 (Xiguan), GB35 (Yangjiao), LI12 (Zhouliao), M-BW-1 (Dingchuan). The depth of needle insertion will be as superficial as 3 mm, and without manual rotation, in order to minimize stimulation of the needle.

All interventions will be performed by the same acupuncturist licensed by the College of Traditional Chinese Medicine Practitioners and Acupuncturists of Ontario (CTCMPAO). Before the acupuncture treatment, appropriate infection control measures will be employed, and different size of single use, sterile, disposable needles in appropriate packages will be available. Participants will be suggested to wear shorts and T-shirts to the lab for their treatments. They will assume a prone position. The skin over points will be swabbed with 70% ethyl alcohol, using an outward rotary motion from the center of the point to the surrounding area to lessen the risk of contamination. No treatment will be taken until the alcohol dries. The acupuncturist will wash his hands immediately before the removal of needles. On withdrawing a needle, a sterile cotton ball will be used to press the skin at the insertion site. If blood is drawn, light pressure will be applied with a clean swab.

The second and third treatment will be on the fifth and third day before the estimated first day of menstruation in each month. The whole process will be repeated at total of nine times over the three months of treatment.

Sample size is calculated from one relatively well designed study. According to this study, the migraine attack frequency each month after treatment in the verum acupuncture group was 4.8 ± 3.8 times, and in the sham acupuncture group 7.8 ± 3.7 times. Based on a power of 0.8 to detect a significant difference (α = .05, two-sided), 32 participants will be required for each group, which is calculated by R software Version 0.96.122 (RStudio, Boston, MA). Allowing for a 20% withdrawal rate, a total of 120 participants will be enrolled with 40 participants in each group.

The analysis will be started once 10 participants have been collected in each group. The statistical significance level will be set at p = .05, and all statistical tests will be two-sided. Factorial analysis of variance (ANOVA) will be used to make comparisons among the three groups. Tukey's post hoc test will be used then to analyze the outcomes of each pair of two groups at each time point. Comparisons within groups for the outcomes at each time point will be done using the one-way ANOVA. All the analyses will be performed using R software Version 0.96.122.

ELIGIBILITY:
Inclusion Criteria:

1. females aged from 18 to 40;
2. a diagnosis of pure menstrual migraine or menstrually related migraine according to the criteria of the International Classification of Headache Disorders III beta version;
3. regular menstrual periods;
4. repeated self-considered MM attacks of at least half a year;
5. no plan to become pregnant or change hormonal treatment during the study; and
6. voluntarily joining this study and providing informed consent.

Exclusion Criteria:

1. difficulties in differentiating migraine from other types of headaches;
2. other primary headaches such as tension-type headache and cluster headache, and secondary headache;
3. lack of time and/or motivation to participate;
4. starting in use of any new kind of migraine prophylactic drugs in the last three months;
5. serious cardiovascular, neurological, or psychiatric diseases according to self-reported medical history;
6. severe bleeding disorder or anticoagulation according to the medical history;
7. a cardiac pacemaker;
8. metal allergy;
9. a severe needle phobia;
10. or if they are pregnant or lactating.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2015-11; Primary Completion 2016-08 (Estimated); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
change from baseline menstrual migraine attack frequency at 9 months | from the date of admission into this study to the date of completion of this study, assessed up to 9 months
  Once the patient is free of headache for 48 hours, a new attack will be considered another headache.

SECONDARY OUTCOMES:
change from baseline number of migraine days at 9 months | from the date of admission into this study to the date of completion of this study, assessed up to 9 months
change from baseline average visual analogue scale (VAS) at 9 months | from the date of admission into this study to the date of completion of this study, assessed up to 9 months
  average visual analogue scale (VAS) for pain ranging from 0 (no pain) to 10 (worst pain) per month
change from baseline total duration period of pain (hours) at 9 months | from the date of admission into this study to the date of completion of this study, assessed up to 9 months
change from baseline number of days with analgesic medication at 9 months | per month, from the date of admission into this study to the date of completion of this study, assessed up to 9 months
change from baseline the absence from work days or school days and/or classes missed at 9 months | from the date of admission into this study to the date of completion of this study, assessed up to 9 months
  the absence from work days or school days and/or classes missed due to menstrual migraine per month

CONTACTS AND LOCATIONS:
Overall Officials: Alan W Salmoni, PhD, Principal Investigator — Western University

REFERENCES:
- [Background] Alecrim-Andrade J, Maciel-Junior JA, Carne X, Severino Vasconcelos GM, Correa-Filho HR. Acupuncture in migraine prevention: a randomized sham controlled study with 6-months posttreatment follow-up. Clin J Pain. 2008 Feb;24(2):98-105. doi: 10.1097/AJP.0b013e3181590d66. PMID 18209514
- [Background] Tfelt-Hansen P, Pascual J, Ramadan N, Dahlof C, D'Amico D, Diener HC, Hansen JM, Lanteri-Minet M, Loder E, McCrory D, Plancade S, Schwedt T; International Headache Society Clinical Trials Subcommittee. Guidelines for controlled trials of drugs in migraine: third edition. A guide for investigators. Cephalalgia. 2012 Jan;32(1):6-38. doi: 10.1177/0333102411417901. No abstract available. PMID 22384463
- [Background] Kong J, Gollub R, Huang T, Polich G, Napadow V, Hui K, Vangel M, Rosen B, Kaptchuk TJ. Acupuncture de qi, from qualitative history to quantitative measurement. J Altern Complement Med. 2007 Dec;13(10):1059-70. doi: 10.1089/acm.2007.0524. PMID 18166116
- [Background] Hu J. Acupuncture treatment of migraine in Germany. J Tradit Chin Med. 1998 Jun;18(2):99-101. PMID 10437224
- [Background] Linde K, Streng A, Jurgens S, Hoppe A, Brinkhaus B, Witt C, Wagenpfeil S, Pfaffenrath V, Hammes MG, Weidenhammer W, Willich SN, Melchart D. Acupuncture for patients with migraine: a randomized controlled trial. JAMA. 2005 May 4;293(17):2118-25. doi: 10.1001/jama.293.17.2118. PMID 15870415
- [Background] Linde M, Fjell A, Carlsson J, Dahlof C. Role of the needling per se in acupuncture as prophylaxis for menstrually related migraine: a randomized placebo-controlled study. Cephalalgia. 2005 Jan;25(1):41-7. doi: 10.1111/j.1468-2982.2004.00803.x. PMID 15606569
- [Background] Sun LH, Li XH, Li WL, Liu L, Ma HL, Liang YL. [Body acupuncture combined with auricular acupressure for menstrual headache: a randomized controlled clinical trial]. Zhen Ci Yan Jiu. 2015 Feb;40(1):70-4. Chinese. PMID 25845225
- [Background] Wang Y, Xue CC, Helme R, Da Costa C, Zheng Z. Acupuncture for Frequent Migraine: A Randomized, Patient/Assessor Blinded, Controlled Trial with One-Year Follow-Up. Evid Based Complement Alternat Med. 2015;2015:920353. doi: 10.1155/2015/920353. Epub 2015 Apr 28. PMID 26060503
- [Background] Jun EM, Chang S, Kang DH, Kim S. Effects of acupressure on dysmenorrhea and skin temperature changes in college students: a non-randomized controlled trial. Int J Nurs Stud. 2007 Aug;44(6):973-81. doi: 10.1016/j.ijnurstu.2006.03.021. Epub 2006 Jun 16. PMID 16782102
- [Background] Lin JA, Wong CS, Lee MS, Ko SC, Chan SM, Chen JJ, Chen TL. Successful treatment of primary dysmenorrhea by collateral meridian acupressure therapy. J Manipulative Physiol Ther. 2010 Jan;33(1):70-5. doi: 10.1016/j.jmpt.2009.11.003. PMID 20114103
- [Background] Diener HC, Kronfeld K, Boewing G, Lungenhausen M, Maier C, Molsberger A, Tegenthoff M, Trampisch HJ, Zenz M, Meinert R; GERAC Migraine Study Group. Efficacy of acupuncture for the prophylaxis of migraine: a multicentre randomised controlled clinical trial. Lancet Neurol. 2006 Apr;5(4):310-6. doi: 10.1016/S1474-4422(06)70382-9. PMID 16545747
- [Derived] Yu X, Salmoni A. Comparison of the Prophylactic Effect Between Acupuncture and Acupressure on Menstrual Migraine: Results of a Pilot Study. J Acupunct Meridian Stud. 2018 Oct;11(5):303-314. doi: 10.1016/j.jams.2018.04.003. Epub 2018 Apr 11. PMID 29654841